

# Official Title: Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029

Date of Protocol: July 14, 2020

NCT Number: NCT04079842



R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



| Protocol/Test Procedure Title | Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029 |
|---|---|
| Lead Investigator | Masimo Corporation 52 Discovery, Irvine, CA 92618 |
| Other Investigators | |
| <b>Expected Start Date</b> | Based on IRB Approval Certification Approval Date |
| Expected End Date | Based on IRB Approval Certification Expiration Date |
| IRB | E&I West Coast Board – IRB00007807 |
| Date Submitted To IRB | |

### **Protocol Test Abstract:**

The objective of this study is to validate the performance of Oxygen Reserve Index (ORi) as computed by the Masimo device in healthy volunteers. The changes in ORi measurements are compared to changes in PaO2 values obtained from arterial blood samples analyzed by a laboratory CO-oximeter reference instrument.

### **APPROVALS**

| Author | Date | Engineering | Date |
|-------------------|------|---------------|------|
| N/A | N/A | N/A | N/A |
| Quality Assurance | Date | Manufacturing | Date |
| N/A | N/A | N/A | N/A |

R-TP - 20088

## Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### STATEMENT OF COMPLIANCE

This document is a protocol for a clinical research study sponsored by Masimo Corporation. The study will be conducted in compliance with all stipulations of this protocol, the conditions of IRB approval, all applicable regulations including 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 812, ISO-14155, and International Conference on Harmonization E6 Good Clinical Practice (ICH GCP).

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study.

#### 1. **PURPOSE**

This test procedure describes the method used to validate the performance of Oxygen Reserve Index (ORi) as measured by the Masimo INVSENSOR00029 sensors connected to the Masimo Radical-7 pulse oximeter and Masimo Root monitor in healthy volunteers. The changes in ORi measurements are compared to changes in PaO2 values obtained from arterial blood samples analyzed by a laboratory CO-oximeter reference instrument.

### Outcome Measure:

This study reports ORi sensitivity and concordance of directional changes in ORi to directional changes in PaO<sub>2</sub> from blood samples (in the range of 100 to 200mmHg).

#### 2. **BACKGROUND**

Masimo Corporation develops non-invasive medical technologies. These devices have applications in the operating room, critical care unit, emergency room, emergency transport vehicles, as well as physician's offices.

An invasive blood sample analyzed by a CO-oximeter reference instrument gives the best measure of arterial oxygen concentration as well as other blood solutes, but cannot measure these parameters continuously and requires skin puncture, arterial line placement and subsequent risk of infection, hematoma, and other physiological damage. Masimo SET and Masimo Rainbow technologies allow real-time, non-invasive monitoring of oxygen saturation (and other blood solutes) and have the potential to improve clinical outcomes while reducing the cost of care and risks to both patients and clinicians associated with arterial and venous punctures.

#### 2.1. **Technology Background**

Pulse oximetry technology is governed by the following principles:

- Oxyhemoglobin (oxygenated blood) and deoxyhemoglobin (non-oxygenated blood) differ in their absorption of red and infrared light (spectrophotometry).
- The amount of arterial blood in tissue changes with arterial pulses (photoplethysmography). Therefore, the amount of light absorbed by the varying quantities of arterial blood changes as well.
- The CO-Oximeter utilizes a sensor with various light-emitting diodes (LEDs) that pass light through the site to a photodiode (detector). See figure below.



- Light Emitting Diodes (LEDs) (2+ wavelengths)
- Detector



# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



### 2.2. Parameter Background

A continuous supply of oxygen is essential for normal cell function. Failure of a patient's oxygen supply to meet metabolic needs is common to all forms of circulatory failure, tissue acidosis, and ultimately mortality. Like all essential commodities for body functions, optimal quantities of oxygen are required. A patient's oxygen status can be largely classified into 3 ranges: Hypoxia (less than normal), Normoxia (normal) and Hyperoxia (more than normal). The three states are typically classified using dissolved oxygen levels in the plasma (PaO<sub>2</sub>), instead of arterial hemoglobin oxygen saturation (SaO<sub>2</sub>), due to sensitivity of PaO<sub>2</sub> in all three states including hyperoxia (unlike SaO<sub>2</sub>). Figure I.<sup>1</sup> shows the three oxygen states based on PaO<sub>2</sub> values along with the relationship between PaO<sub>2</sub> and SpO<sub>2</sub> (which is a proxy for SaO<sub>2</sub>)

### OxyHemoglobin Dissociation Curve



Figure 1: The oxygen dissociation curve with the three oxygen states

Currently, in order for clinicians to monitor a patient's oxygen status, both continuously and non-invasively, they utilize a pulse oximeter to obtain  $SpO_2$  (a proxy for  $SaO_2$ ) levels. However,  $SpO_2$  is sensitive in the normoxic and hypoxic regions and largely remains flat in the hyperoxic region (Figure 1) clinicians generally resort to invasive blood draws to obtain  $PaO_2$  values which provide oxygen status within the hyperoxic zone. This method has multiple drawbacks such as intermittent samples to potential delay between time of blood draw to the time when the  $PaO_2$  value is obtained through blood gas machines.

The ORi Parameter may help provide clinicians with a convenient noninvasive method for monitoring oxygenation status in the moderate hyperoxic range, that may be used in conjunction with SpO2 and reference  $PaO_2$  measurements. While not a direct measurement of  $PaO_2$ , ORi is intended to provide a continuous and non-invasive directional trending index which reflects directional changes in oxygenation. The concordance of directional changes to  $PaO_2$  from blood samples is used to validate the ability of ORi to monitor oxygenation status in the moderate hyperoxic range (in the range of 100 to 200mmHg).

<sup>&</sup>lt;sup>1</sup> Martin, L. (1999). All you really need to know to interpret arterial blood gases, Page 73, Lippincott Williams & Wilkins.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



### 2.3 Investigational Study Devices

The investigational devices to be used in this study are the Masimo INVSENSOR00029 rainbow disposable sensor, Masimo Radical-7 Pulse CO-Oximeter, and Masimo Root Patient Monitoring and Connectivity Platform. The investigational sensor is equivalent to the FDA cleared sensors with regard to intended use on the surface of the skin, the choice of materials, biocompatibility, manufacturing process and risk of exposure to the subject to any energy or light source. They do not pose any additional risk to patients as compared to the similar FDA cleared sensors. The Masimo Root Patient Monitoring Platform is an FDA-cleared patient monitoring and connectivity platform that offers rainbow and Masimo SET measurements with other parameters in an integrated platform. With docking capabilities for the Radical-7° handheld monitor and multiple networking/connectivity options, Root integrates multiple streams of data into one display monitor. The Masimo Radical-7 pulse oximeter is an FDA-cleared noninvasive monitoring platform featuring Masimo SET Measure-through Motion and Low Perfusion™ pulse oximetry with the option to measure multiple additional blood constituents and physiologic parameters.

<sup>&</sup>lt;sup>2</sup> D. S. Martin and M. P. W. Grocott III., Oxygen therapy in anaesthesia: the yin and yang of O2 Br. J. Anaesth. (2013) 111 (6): 867-871 doi:10.1093/bja/aet291

<sup>&</sup>lt;sup>2</sup> Habre W1, Peták F2. Perioperative use of oxygen: variabilities across age. Br J Anaesth. 2014 Dec;113 Suppl 2:ii26-ii36. doi: 10.1093/bja/aeu380

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### 3. REFERENCE

Consent To Be A Research Subject Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029

Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029 Case Report Form (CRF)

Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029 Healthy Volunteers Needed Advertisement

Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029 Recruitment

Script

Health Assessment Questionnaire Health Assessment Questionnaire Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029

- Confidentiality Agreement
Volunteer payment form
Informed Consent Process
Clinical Study Request Form (CSRF)
Post Care Instructions

#### 4. LOCATION

Masimo Corporation

**Clinical Laboratory** 

52 Discovery

Irvine, CA 92618



### 5. STUDY POPULATION

### 5.1. Inclusion Criteria

- Subject is 18-50 years of age.
- Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
- Hemoglobin value is greater than or equal to 11 g/dL.
- Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
- CO value  $\leq$  2.0% FCOHb.
- Subject has a physical status of ASA I or II (American Society of Anesthesiology Class 1; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
- Blood Pressure: (Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥50 mmHg), and if blood pressure is lower than 100/60 subject passes an orthostatic blood pressure test
- Subject is able to read and communicate in English and understands the study and risks involved.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



- 5.2. **Exclusion Criteria** (\*= Per physician discretion)
  - Subject is pregnant.
  - Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
  - Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
  - Subject smokes one pack of cigarettes or more in one week, and/or the equivalent of e-cigarette liquid, and smokers are not being recruited as indicated in the CSRF.
  - Subject has open wounds, inflamed tattoos or piercings and/or any visible healing wounds that a
    medical professional renders them at an increased risk for participation.\*
  - Subject has known drug or alcohol abuse or uses recreational drugs.
  - Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
  - Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
  - Subject has any history of a stroke, myocardial infarction, seizures or heart attack.
  - Subject who has taken anticoagulant medications within the last 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDS).
  - Subject has donated blood within the past 4 weeks.
  - Subject has any chronic bleeding disorder (i.e. hemophilia)
  - Subject has any symptomatic cardiac dysrhythmia (i.e. atrial fibrillation) and has not received clearance from their physician to participate.
  - Subject has Wolff-Parkinson-White Syndrome or Stokes Adams syndrome.
  - Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subjects' level of consciousness.
  - Subject has taken opioid pain medication within 24 hours of start of study.
  - Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
  - Subject is taking medications known to treat any type of infectious disease.\*
  - Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
  - Subject has had invasive surgery within the past year- including but not limited to major dental surgery\*, appendix\*, plastic surgery\*.
  - Subject has had invasive surgery within the past year- including but not limited to gallbladder, major fracture repairs (involving plates/ screws), jaw surgery, urinary tract surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
  - Subject has symptoms of congestion, head cold, flu or other illnesses.
  - Subject is claustrophobic and/or has generalized anxiety disorder.
  - Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
  - Subject has any cancer or history of cancer (not including skin cancer).\*
  - Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
  - Subject is allergic to lidocaine, latex, adhesives, or plastic.
  - Subject has a heart condition, insulin-dependent Diabetes, or uncontrolled hypertension.
  - Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the past 6 months.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



- Subject intends to participate in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involved an arterial line.
- Subject has any medical condition which in the judgement of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator/study staff).

### 5.3. Withdrawal of subjects

Subjects must be withdrawn under the following circumstances:

- 5.3.1 The subject withdraws consent.
- 5.3.2 Discretion of investigator, for example:
  - The investigator feels that the subject is too money motivated.
  - The investigator feels that the subject does not fully comprehend and understand the consent form.
  - The subject is ill-mannered and/or shows aggressive behavior towards study staff.
  - Malfunction of the device for greater than 30 minutes that prevents accurate collection of optical data.
  - Subject displays or communicates signs of discomfort or distress so that the study may not be continued.

### 5.4. Replacement of subjects

In case a subject is withdrawn from the study, another subject may be recruited.

### 6. EQUIPMENT AND MATERIALS

Equipment and Materials: All lab analyzers and equipment will be maintained per manufacturer specifications and all study personnel will be trained on the use of relevant equipment. Equivalent equipment and materials to those listed below may be used.

### Safety Equipment (FDA-Cleared)

- Blood pressure monitoring system
- Electrocardiogram (ECG)
- Masimo Pulse Oximeters (Radical-7) for subject safety monitoring
- Pulse oximeter sensors and cables (Masimo SET, Masimo rainbow)
- Masimo Patient Monitoring Platform (Root®)- for subject safety monitoring
- Medical-grade Oxygen tank and mask
- Crash cart

### **Test Devices**

- Masimo INVSENSOR00029 sensor Investigational
- Masimo Patient Monitoring Patform (Root®)
- Masimo Pulse Oximeters (Radical-7)

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



### Research Equipment

- Laboratory co-oximeters/blood analyzers

### 7. PROCEDURE

### 7.1 SCHEDULE OF ACTIVITIES



R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### 7.2. RECRUITMENT AND PRESCREENING

Subjects will be recruited using IRB-approved advertisements. Subjects may be referred to the study by previous subjects. Subjects are contacted via phone call to conduct a prescreening interview to determine their initial eligibility for the study. Potential eligible subjects are scheduled for a study visit to the clinical laboratory.

#### 7.3 **CONSENTING AND SCREENING**

Study staff will discuss the informed consent process and the study with the potential subjects. The subjects will be provided with enough time to read and understand the informed consent document and their questions will be answered by study staff prior to the subject signing the informed consent form. No study related activities will be conducted until consent is signed.

Subjects will be asked to provide a copy of their valid government photo ID and/or Social Security Number (SSN) card to verify subject identity. The copies of these forms of identification will be stored along with the subject's consent. The confidentiality and retention of these documents will be protected to the extent provided and required by law.

Subjects will be asked a brief series of health questions to ensure their eligibility for this study. Subjects who do not meet the inclusion and exclusion criteria will not be eligible to participate in the study.



In addition, a medical history will be recorded after the initial screening questionnaire.

Pre-procedure vital signs will be recorded for subject safety monitoring. Spikes in blood pressure and heart rate can be expected during line placement, needle sticks, blood draws etc. and may also be attributed to anxiety/nervousness relating to a new environment. Only the initial recorded blood pressure and/or heart rate determines a subject's qualification for the study.

A physician will perform an orthostatic blood pressure test on subjects with an initial blood pressure

The orthostatic blood pressure test will start with the physician taking the subject's blood pressure while they are lying in supine position. The subject will then stand up for 30 seconds and a second blood pressure measurement will be taken. The subject's blood pressure will need to stay to meet inclusion criteria for the study.

Female subjects will be required to take a pregnancy test. Results will be noted in study documentation. If the pregnancy test is positive, the subject will be notified and removed from the study.



Subjects may have a blanket placed on them for their comfort.

Subjects may be offered a snack (e.g., granola bar) and/or beverage (e.g., water, juice) due to the amount of time their involvement in this study may take.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



### 7.4. PROCEDURES

If accepted into the study, standard hospital-type monitors will be placed on the subject, including ECG, blood pressure, and a reference pulse oximeter for safety monitoring by medical staff.

Local anesthetics such as lidocaine, ethyl chloride spray, or Pain Ease skin refrigerant spray may be used in the event that an IV is placed to numb the site. Subjects will be given the option to have lidocaine or numbing spray be used during IV placement for the purpose of making catheter placement more comfortable for the subjects.

, sensors will be placed on the required sensor sites.

The timing of all the blood draws will be entered into the data collection software.

If at any point the subject is uncomfortable with the study, the study will be stopped.

### 7.5. END OF STUDY PROCEDURE

At the conclusion of the procedure, the sensors/devices, IV(s), will be removed and the subject will be allowed to leave after medical personnel determine it is safe to do so.

Study staff may take to verify the subjects blood values are within normal range (eg. pH, Glucose, etc.)

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



All subjects will be encouraged to remain in the study area until they feel fit to leave; subjects should feel safe and able before returning to work directly after participation in the study.

Subjects will be given instructions on wound care. All subjects will be instructed to contact the principal investigator or study staff in the event of any potential complication.

Subjects will be paid for their time.

After the study has ended subjects will be offered a snack (e.g., Granola bar) and something to drink (e.g., water or juice). Subjects are asked to consume food and/or liquid prior to leaving the clinical lab area for their safety due to study procedures such as blood removal and subjects may also be asked to wait in the clinical lab or lobby waiting area for an additional 30 minutes (estimate) before leaving to allow for their body to continue adjusting after the study has completed.

### 7.6. RE-CONTACTING SUBJECTS

If the subject fails to provide proper documentation on their individual consent form for any study, Masimo has the right to re-contact the subject and ask them to return to the clinical lab in order to properly complete the consent form or subject bill of rights. Subject will be compensated for travel.

The subject will also fill out other study documents. These documents aid in the collection of data, tracking subject count, etc. If the subject fails to provide proper documentation on other documents, Masimo has the right to re-contact the subject and ask them to return to the clinical lab in order to properly complete these documents if seen as necessary by study staff.

The subject will be re-contacted via phone or email and be asked to return as soon as possible.

| 8. | ACCEPTANCE ( | CRITERIA (JUSTIFY | <b>IF NOT</b> | APPLICABLE) |
|----|--------------|-------------------|---------------|-------------|

9. SAMPLE SIZE JUSTIFICATION



### 10. DATA ANALYSIS PROCEDURE TO BE USED

### **EXCLUSION CRITERIA FOR DATA ANALYSIS**

In order to ensure the validity of the measurements, each ORI/PaO2 data pair was evaluated through the following criteria to remove samples that could be erroneous due to various reasons such as Reference Errors, User Errors, or ORI monitoring system Quality Checks as listed below

- 1. Reference Errors: Samples reported with an exception (e.g., "Error Codes from reference machine") from reference machine are discarded for data analysis, since the PaO2 measurement may not be reliable or will not be available.
- 2. ORI monitoring system error: Samples reported with ORI system exception are discarded for data analysis, since the ORi value may not be available or reliable.
- 3. Incomplete study: Data from subjects who did not go through the full protocol are excluded from data analysis

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



- 4. For a given FiO2 level, each of the discarded, since the sampling time difference may result in the data not being reflective of one another resulting in the erroneous inclusion of the PaO2 reference for data analysis. Also PaO2 blood draws with values with differences are discarded for data analysis, as the difference may be reflective of an erroneous or inconsistent PaO2 reference.
- 5. Exclusion Criteria for PaO2 levels outside ORI sensitive region (100 to 200 mmHg)
  - a. PaO2 values below 100 mmHg and above 200 mmHg are discarded for data analysis, as the focus of the study is the validation of ORi in the moderate hyperoxic range (of 100 to 200 mmHg PaO2).
- 6. Samples with  $|\Delta PaO2|$  or  $|\Delta ORI|$  are excluded for data analysis of the sensitivity, specificity or concordance computation, since these changes are not considered significant reflections of changes in oxygen status based upon the repeatability and reproducibility analysis described below.

 $\Delta$ PaO2 and  $\Delta$ ORI were computed by taking the difference of all ORI and PaO2 readings from the study with this chosen PaO2 threshold level.

 $\Delta$ PaO2 and  $\Delta$ ORI computation are defined as:

 $\Delta PaO2 = PaO2(t) - PaO2(tref)$ 

 $\Delta ORI = ORI(t) - ORI(tref)$ 

where 'tref' is the time of the sample closest to PaO2threshold in a window

't' represents all other time synchronized ORI/PaO2 data pair from the study



Specificity, sensitivity and concordance will be computed for changes in ORi with respect to changes in PaO2 as described below:

#### ΔPaO<sub>2</sub> vs ΔORI

ΔPaO<sub>2</sub> and ΔORI are defined below.

$$\Delta PaO_2 = PaO_2(t) - PaO_2(t_{ref})$$

where  $t_{ref}$  is the time of the sample closest to  $PaO_{2threshold}$  in a window is used as it is not possible to draw a blood sample at the exact desired value of  $PaO_{2\,threshold}$ .  $PaO_{2\,can}$  be any value from 110 to 190 in steps of 10mmHg (see footnote) to cover the range of 100 to 200mmHg.

 $\Delta ORI = ORI(t) - ORI(t_{ref})$ 

Samples with  $\Delta PaO_2$  of  $\pm$  10 mmHg are ignored (see footnote<sup>+</sup>).

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



- 1) As per Figure 2, specificity is defined as Specificity = N1 / (N1 + N4)
- 2) As per Figure 2, sensitivity is defined as Sensitivity = N3 / (N2 + N3)
- 3) As per Figure 2, concordance is defined as Concordance = (N1 + N3) / (N1 + N2 + N3 + N4)

The relationship between Concordance, Specificity and Sensitivity is as shown below.

Let 
$$N = (N1 + N2 + N3 + N4)$$

Concordance  $= \frac{N1}{N} + \frac{N3}{N}$ 
 $= \frac{N1 (N1+N4)}{N (N1+N4)} + \frac{N3 (N2+N3)}{N (N2+N3)}$ 
 $= \frac{N1+N4}{N} * Specificity + \frac{N2+N3}{N} * Sensitivity$ 

Concordance =  $\alpha * Specificity + (1 - \alpha) * Sensitivity$ where  $0 \le \alpha \le 1$ .



Figure 2: Specificity and Sensitivity Illustration for  $\Delta PaO_2$  vs  $\Delta ORI$ 

<sup>&</sup>lt;sup>5</sup> Bedford, Robert F. MD, (1978), Long-term radial artery cannulation: effects on subsequent vessel function, *Critical Care Medicine*, *6* (1), 1-71.

<sup>&</sup>lt;sup>5</sup> Slogoff S, Keats AS, Arlund C, (1983), On the safety of radial artery cannulation, *Anesthesiology*, *59* (1), 42-47.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### 11. ADVERSE EVENTS

**Definitions:** 

<u>Adverse event</u>: Any untoward medical occurrence in a subjects, users or other persons, whether or not related to the medical device under study.

<u>Device-related adverse event</u>: Adverse event related to, associated with, or caused by, the use of a medical device under study, including but not limited to events that may have been attributed to the device because of device failure or malfunction, improper or inadequate design, manufacture or user error.

<u>Device deficiency</u>: Inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety or performance. Device deficiencies include malfunctions, use errors and inadequate labeling. Device deficiencies will be reported according to department procedures.

<u>Serious adverse event</u>: Adverse event that: a) led to death, b) led to serious deterioration in the health of the subject, that resulted in: (i) a life-threatening illness or injury, (ii) a persistent or significant impairment of a body structure or a body function, (iii) in-patient or prolonged hospitalization, or (iv) medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function, or c) led to fetal distress, fetal death or a congenital abnormality or birth defect. NOTE: Planned hospitalization for a pre-existing condition, or a procedure required by the clinical investigational plan, without serious deterioration in health, is not considered a serious adverse event.

All adverse events, including inter-current illnesses will be reported and documented as described below.

#### 11.1 Adverse Events

All adverse events that occur during the study shall be recorded on the Case Report Form even if the investigator/study staff assesses the adverse event as unlikely to be causally related to the test device or study procedures.

#### 11.2 Serious Adverse Events

The investigator/study staff shall promptly report both serious adverse events and unanticipated adverse device effects to the sponsor within 48 hours. All serious adverse events will also be reported to the IRB per IRB reporting requirements.

At the time of discharge from the study, any unresolved serious adverse event(s) will be followed up by the investigator/study staff until the event(s) are resolved, stabilized or the patient is lost to follow-up or the adverse event is otherwise explained. The investigator/study staff will also instruct the subject to report any subsequent events occurring in the next 30 days, which the subject or the subject's physician believes might reasonably be regarded as caused by or have a reasonable possibility of being caused by the test device or procedures involved in the study.

### 11.3 Unanticipated Problems

Any unanticipated problem involving subjects will be reported to the IRB, such as protocol violations or deviations as required by the IRB reporting procedures.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### 12. SUPPORTING DOCUMENTATION AND OPERATIONAL CONSIDERATIONS

- 12.1 Measures Taken to Protect the Rights and Welfare of Subjects
  - 12.1.1 All subjects will be monitored closely throughout the study. There will be an ACLS certified medical doctor present in the study area throughout the study.
  - 12.1.2 The following measures will be taken to ensure the confidentiality of the subjects:
    - 12.1.2.1 A code (identification) number for each subject will be kept on file.
    - 12.1.2.2 Only their corresponding identification number will identify subjects.
    - 12.1.2.3 Access to identifying documents (IC, SSN, photo ID) and data will only be made to the principal investigators in the study and study staff.
    - 12.1.2.4 The confidentiality and retention of these documents will be protected to the extent provided and required by the law.

### 12.2 Vulnerable Populations

12.2.1 Employees are considered to be a vulnerable population.

Participation is not a condition of employment. There will be no repercussions in the workplace in the case that the employee refuses to participate in the study or withdraws at any point during the study. Neither supervisors nor superiors will be involved in the recruitment of employees for participation in the study.

12.2.2 Economically disadvantaged or unemployed and educationally disadvantaged.

Reasonable compensation will be provided for economically disadvantaged subjects to eliminate possibility of undue influence due to financial incentive. Educationally disadvantaged subjects will be provided ample time to ask questions and comprehend information.

### 12.3 Documents and Database

| 12.3.1 | .1 Documents will be kept a grant after the sp longer being made. If destroyed, these documents will be company used for destroying medical and clinical data. | ecific product/tested for is no eshredded and done by a certified |
|---|---|---|

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



#### 13. DEVICE ACCOUNTABILITY

### 13.1 Receipt of Study Device

Upon receipt of the study device supplies, an inventory must be performed and the device accountability log filled out and signed by the person accepting the shipment. It is important that the designated study staff counts and verifies that the shipment contains all the items noted in the shipment inventory. Any damaged or unusable study devices in a given shipment will be documented in the study files.

### 13.2 Use of Study Device

Use of devices and sensors will be documented on Case Report Forms for each subject.

### 13.3 Return or Destruction of Study Device

At the completion of the study, there will be a final reconciliation of study devices and sensors shipped, devices/sensors used, and devices/sensors remaining. This reconciliation will be logged on the device accountability log. Any discrepancies noted will be investigated, resolved, and documented prior to return or destruction of unused study devices. Devices destroyed on site will only be upon written instruction from the sponsor and will be documented in the study files.

#### 14. RISKS AND BENEFITS

- 14.1 Benefits: There will be no benefit to the subject. Other possible benefits would be to society as a whole. Evaluation of the accuracy of this new device could enable healthcare workers to more appropriately treat potentially life threatening conditions.
- 14.2 Device Risks: The noninvasive devices used in this study are similar in technology and design to some commercially available pulse oximeters and other non-invasive devices and hence have the same risks. Pulse oximeters and other non-invasive devices are commonly used and are considered to be minimal risk. There is an extremely small risk of damage to the subject's fingers, or other locations where sensors are placed, from the device including temporary skin irritation or discomfort associated with exposure to the sensor as well as potential temporary mechanical irritation or discomfort. There is a remote, yet possible, risk of a burn from the sensor. In the case of a sensor burn there is the potential for permanent skin damage (scar/discoloration).
- 14.3 Venous Cannulation Risks: swelling, infection, infiltration of fluids/ blood into area surrounding IV, bruising, hematoma, lightheadedness, fainting, feeling flush/warm, feeling nauseated, throwing up, sudden drop in blood pressure/sudden increase in blood pressure, sudden drop in heart rate/sudden increase in heart rate, tingling sensation of face, arms and/or legs, sweating, mouth dryness, damage to the blood vessel and surrounding nerves or tissue.
- 14.4 Arterial Cannulation risks: decreased blood supply, blood clot, embolization, infection, hematoma, damage to the blood vessel and surrounding nerves, tendons or tissue; loss of feeling in hand and/or arm and even the loss of hand due to rare complications of the study.
- 14.5 Blood Draw risks: discomfort is generally associated with needle puncture. The most common complications associated with blood draws and capillary sticks are hematomas or bruising. All blood draws will be performed by qualified personnel. An ACLS certified physician will be in attendance throughout the entire procedure, and the study will be completed under their general supervision.

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



Other anticipated adverse events that may occur, include but are not limited to: vasovagal (passing out/fainting), infection to the skin or area right below the skin, lightheadedness, feeling flush/ warm, feeling nauseated, throwing up, seizures, sudden drop in blood pressure/ sudden increase in blood pressure, sudden drop in heart rate/ sudden increase in heart rate, tingling sensation of face/arms and/or sweating, and mouth dryness. These anticipated adverse events are expected to be temporary.

- 14.6 Risk From Oxygen Administration: It is expected that some people may experience feelings of claustrophobia or anxiousness from wearing a mouthpiece and/or mask. There are no additional risks associated with high oxygen/oxygen administration for less than 24 hours as long as subjects do not have any cardiac conditions, COPD or any other lung diseases. Subjects' answers on the health questionnaire will help the medical staff decide if they can safely participate in this study; subjects are encouraged to let the study staff know if they have any concerns.
- 14.8 Risk from Inflicted Knowledge: The risk of inflicted medical knowledge to subjects is negligible since we de-identify all associated sample information including those relevant to our clinical and engineering parameter studies. The monitoring and test results are not examined for diagnostic purposes and do not reflect an attempt to ascertain any subject's medical condition. The attending physician's role during this study is to ensure the safety of the subject during the study. Subjects are informed that these are not diagnostic tools, if observations are made using FDA cleared devices we will refer them to their primary care physician.
- 14.9 Risk From Loss of Confidentiality: Masimo upholds the highest standards to protect hard and electronic data however, a complete promise for confidentiality cannot be guaranteed due to unforeseeable events.
- 14.10 Risk From Additional Testing:
  - 14.10.1 During the conduct of the study, it is possible, but not likely, that someone could become exposed to the sample of blood drawn from the subject through an inadvertent needle stick or by contact with an open cut. In such circumstances, it will be important to the exposed individual to know whether the blood to which he or she was exposed contained Hepatitis B virus (HBV), Human immunodeficiency virus (HIV), or Hepatitis C virus (HCV) and additional testing of the sample will be performed.
  - 14.10.2 Within the consent, subjects will agree to permit the company to test the blood sample (or samples) by signing the consent. The test results will be maintained as confidential and will only be used by healthcare professionals for the diagnosis and treatment of the exposed individual as appropriate.
  - 14.10.3 In the case that Masimo needs to contact a subject regarding additional testing they will be contacted by a Masimo employee and medical personnel can be available for further counsel if requested.
  - 14.10.4 The cost for the initial testing and compensation for their time/travel to the testing facility will be the only things paid for by Masimo.
- 14.11 Lidocaine (injection) Risks: Insertion of the Lidocaine may be discomforting and can feel like a slight pinch along with a warm/burning sensation. Other anticipated adverse events that may occur,

R-TP - 20088

# Oxygen Reserve Index (ORi) Expanded Data Set Validation of INVSENSOR00029



include but are not limited to: Flushing or redness of the skin, itching skin, small red or purple spots on the skin, unusually warm skin, bruising, bleeding at the application site, and swelling, feeling nauseated, dizziness, low blood pressure, and/or tremors. These adverse events are expected to be temporary.

Although not common, it is also possible to have an allergic reaction to injectable lidocaine (e.g. seizures). Subjects should not take part in this study if they are allergic to lidocaine injection or other types of numbing medicine, or if they have a heart rhythm disorder such as Wolff-Parkinson-White Syndrome or Stokes-Adams syndrome. Subjects are instructed to tell the study staff right away if they experience hives; difficulty breathing; swelling of your face, lips, tongue or throat.

14.12 Ethyl Chloride (Lidocaine Spray): Ethyl Chloride is a topical anesthetic which is used to prevent pain by cooling the skin. Although unlikely, the anticipated adverse events that may occur, include but are not limited to: changes in skin color (i.e. Flushing or redness of the skin), delayed wound healing, rash, itching and swelling. These adverse events are expected to be temporary.

#### 15. EMERGENCY RESPONSE PLAN FOR MEDICAL EMERGENCIES

The physician and nurse present during the study will be ACLS certified and will respond to any medical emergency involving a subject with the ACLS approved protocol for intervention. A crash cart is on site and full emergency services are within 3 miles.

### 16. MONITORING PLAN

A separate document for the study monitoring plan will be developed and followed to ensure subject safety and GCP compliance.

### 17. PROTOCOL DEVIATIONS AND AMENDMENTS

Deviations to the protocol will be documented on the Case Report Form or a separate document. Protocol deviations will be reported to the sponsor and IRB per IRB reporting guidelines.

Modifications to the protocol, informed consent materials, recruitment materials, or any other materials provided to subjects must be reviewed and approved by the IRB.